CLINICAL TRIAL: NCT03556748
Title: Effect of Whole-body Electromyostimulation Combined With Individualized Nutritional Support on Patients With Hematological Malignancies
Brief Title: WB-EMS and Nutrition in Patients With Hematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMS Nutr hemato onko
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Hematologic Diseases; Cachexia; Cancer; Leukemia; Myeloma; Lymphoma; Cancer
Keywords: hematological malignancies; leukemia; myeloma; lymphoma; exercise; nutrition; protein; WB-EMS; whole-body electromyostimulation
MeSH Terms: conditions — Hematologic Diseases; Cachexia; Neoplasms; Leukemia; Neoplasms, Plasma Cell; Lymphoma; Hematologic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: WB-EMS training is performed 2x/week for 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): usual care" control group receives individualized nutritional support (dietary advices: daily protein intake 1.2-1.5 g/kg bodyweight),
  active exercise therapy is optionally provided (bicycle ergometers at room) during the in-Patient stay
- WB-EMS group (Experimental): physical exercise group regular WB-EMS training (2 EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake 1.2-1.5 g/kg bodyweight)
  active exercise therapy is optionally provided (bicycle ergometers at room) during the in-Patient stay
  Interventions: Other: whole-body electromyostimulation

INTERVENTIONS:
Other: whole-body electromyostimulation — WB-EMS training is performed 2x/week for a total of 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
  Arms: WB-EMS group

SUMMARY:
This study evaluates the effects of a whole-body electromyostimulation (WB-EMS) training combined with individualized nutritional support on skeletal muscle mass, body composition, muscle strength/function, quality of life, fatigue, pain and gastrointestinal symptoms in patients with hematological malignancies 4-6 weeks before and 4-6 weeks after undergoing stem cell Transplantation. Within this context, this study also investigates the effect of the nutrition and exercise intervention on the period of hospitalization, period of White blood cell recovery and frequency and severity of complications (mucositis, Graft-versus-Host-Disease, infections) after stem cell Transplantation as consequences of the therapeutic immune Suppression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with hematological malignancies with an indication for stem cell Transplantation
* Interval until Transplantation: 6 weeks
* ECOG Status 0-2

Exclusion Criteria:

* patients with serious osteolytic lesions and increased risk of fall
* simultaneous participation in other nutritional or exercise intervention Trials or in the past 6 months
* acute cardiovascular events
* use of anabolic medications
* epilepsy
* severe neurological diseases
* skin lesions in the area of electrodes
* energy active metals in body
* acute vein thrombosis
* rheumatic diseases
* pregnant and nursing women
* psychiatric disorders with doubts about legal and cognitive capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mass | 12 weeks
  Skeletal muscle mass assessed by bioelectrical impedance analysis (in kg)

SECONDARY OUTCOMES:
Physical function - Isometric muscle strength | 12 weeks
  Hand grip strength assessed by hand dynamometer (in kg)
Cardiorespiratory Fitness | 12 weeks
  VO2max assessed by spirometry
Patient-reported Quality of Life (QoL) | 12 weeks
  EORTC QLQ - C30 questionnaire
Patient-reported Fatigue | 12 weeks
  FACIT-Fatigue scale
Depression/Anxiety | 12 weeks
  Hospital Anxiety and Depression Scale
Inflammatory blood markers | 12 weeks
  Blood collection and analysis (Albumin, CRP, Cytokines)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany